CLINICAL TRIAL: NCT03559894
Title: Severe and Transient Hypoxemia During Selective Intra-arterial Chemotherapy for Retinoblastoma in Children: Evaluation of the Right-sided Heart Function.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Christian Kern (Other)
Responsible Party: Sponsor-Investigator, Christian Kern, Professor, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Other Study IDs: 2017-01539
Record Dates: First submitted 2017-10-19; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Trans-thoracic echocardiography — Trans-thoracic echocardiography

SUMMARY:
Children having selective ophthalmic artery chemotherapy for retinoblastoma under general anaesthesia may experience troubles during the procedure. The troubles are transient, may be severe and include hypoxemia, hypotension and bradycardia. All children having such trouble always fully recovered without any sequelae or prolonged length of stay. The investigators suspect that these phenomenons are caused by transient pulmonary hypertension.The objective is to see whether transient pulmonary hypertension and right-sided heart failure is present during theses phenomenon by trans-thoracic echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Retinoblastoma requiring selective ophthalmic artery chemotherapy under general anaesthesia

Exclusion Criteria:

* Obesity
* pre-existing significant heart or pulmonary disease.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children 0 to 6 years old having selective ophthalmic artery chemotherapy for retinoblastoma under general anaesthesia are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Identification of pulmonary hypertension and/or right-sided heart failure (systolic arterial pulmonary pressure and visual function of the right ventricle is measured) | Perioperative.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Phillips TJ, McGuirk SP, Chahal HK, Kingston J, Robertson F, Brew S, Roebuck D, Hungerford JL, Herod J. Autonomic cardio-respiratory reflex reactions and superselective ophthalmic arterial chemotherapy for retinoblastoma. Paediatr Anaesth. 2013 Oct;23(10):940-5. doi: 10.1111/pan.12162. Epub 2013 May 13. PMID 23668238
- [Result] Kato MA, Green N, O'Connell K, Till SD, Kramer DJ, Al-Khelaifi M, Han JH, Pryor KO, Gobin YP, Proekt A. A retrospective analysis of severe intraoperative respiratory compliance changes during ophthalmic arterial chemosurgery for retinoblastoma. Paediatr Anaesth. 2015 Jun;25(6):595-602. doi: 10.1111/pan.12603. Epub 2015 Jan 7. PMID 25565164
- [Result] Scharoun JH, Han JH, Gobin YP. Anesthesia for Ophthalmic Artery Chemosurgery. Anesthesiology. 2017 Jan;126(1):165-172. doi: 10.1097/ALN.0000000000001381. No abstract available. PMID 27748655
- [Result] Monroy JE, Orbach DB, VanderVeen D. Complications of intra-arterial chemotherapy for retinoblastoma. Semin Ophthalmol. 2014 Sep-Nov;29(5-6):429-33. doi: 10.3109/08820538.2014.959188. PMID 25325870
- [Result] Schaller B, Cornelius JF, Prabhakar H, Koerbel A, Gnanalingham K, Sandu N, Ottaviani G, Filis A, Buchfelder M; Trigemino-Cardiac Reflex Examination Group (TCREG). The trigemino-cardiac reflex: an update of the current knowledge. J Neurosurg Anesthesiol. 2009 Jul;21(3):187-95. doi: 10.1097/ANA.0b013e3181a2bf22. PMID 19542994